CLINICAL TRIAL: NCT06776289
Title: Endodontic Microsurgery With and Without Platelet-Rich Fibrin
Brief Title: Endodontic Microsurgery
Acronym: EMS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mark Schachman (Other)
Responsible Party: Sponsor-Investigator, Mark Schachman, Post Graduate Program Director in Endodontics, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 95694
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Apical Periodontitis
Keywords: endo; endodontic; microsurgery; apicoectomy; apico; prf; platelet rich fibrin
MeSH Terms: conditions — Periapical Periodontitis; Endometriosis

STUDY DESIGN:
Intervention Model Description: Participants will be placed in group A or group B. Group A will have endodontic microsurgery without the use of PRF and group B will have endodontic microsurgery with the use of PRF.
Who Masked: Outcomes Assessor
Masking Description: Oral Radiologist assessing healing will not be aware if the patient had received PRF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microsurgery with Platelet Rich Fibrin (Experimental): Patents will have a blood draw completed so that PRF can be made. Endodontic microsurgery will then be completed. Prior to closing the flap, PRF will be placed in the osteotomy.
  Interventions: Biological: Platelet rich fibrin
- Microsurgery Alone (No Intervention): Endodontic microsurgery will be completed without PRF. The osteotomy will remain empty as per standard procedure.

INTERVENTIONS:
Biological: Platelet rich fibrin — Platelet rich fibrin will be used to fill an osteotomy after endodontic microsurgery is completed.
  Arms: Microsurgery with Platelet Rich Fibrin

SUMMARY:
Current literature on platelet rich fibrin (PRF) use in apicoectomies, also known as endodontic microsurgery, is sparse. PRF use in oral surgery or periodontal surgery has been more thoroughly researched. Whether it is able to reduce post-op pain or if it improves success rate in endodontic microsurgery is not well known. It is also not well known if it will be able to increase the rate of healing. This study will evaluate the success of endodontic microsurgery with and without PRF.

DETAILED DESCRIPTION:
Periradicular surgery is an endodontic procedure comprising of surgical access to the periapical area to perform direct periradicular curettage, root-end resection, root-end preparation and filling. In situations where the outcome of primary root canal treatment is not sufficient, nonsurgical retreatment is considered the option of choice. Surgical endodontic treatment is usually employed to manage apical periodontitis when the orthograde approach (root canal treatment or retreatment) to the apical root anatomy (and infection) is irretrievably obstructed.

However, If the existing root canal anatomy cannot be successfully explored and instrumented with the radiographic presence of apical periodontitis, nonsurgical retreatment has been reported to be as low as low as 40%. In addition, a variety of tooth-related factors may necessitate surgical retreatment, including complicated root canal anatomy, the pathophysiology of the apical pathosis, extreme root curvatures, severe root canal alterations caused during treatment, non-removable root filling materials, existing posts at great risk for retreatment, and root fractures as well as perforations, resorptions, or root fractures. Furthermore, a surgical approach may be indicated when the periradicular tissues require direct visualization, debridement, excision, biopsy or management due to biomechanical failures.

Yan et al. found that the use of concentrated growth factors may influence the outcome of endodontic microsurgery. A systematic review by Mehta found that the use of platelet aggregates, such as PRF gave a favorable effect on the healing of apico-marginal defects, the research suggests that more studies are needed on the healing outcomes of endodontic microsurgery with PRF.

PRF has been widely used in regenerative dentistry, periodontics, and oral surgery with varying degrees of success. It is made through centrifugation of peripheral blood with the resulting centrifuged product is a solid fibrin clot sandwiched between the supernatant and blood cells. The matrix of the solid fibrin clot is a matrix consisting of platelets, leukocytes, a variety of growth factors, and cytokines as well as high biocompatibility due to its autologous source.

In this study patients will receive endodontic microsurgery with one group having the osteotomy filled with PRF prior to closure and another group having surgery completed without the use of PRF. Healing will be evaluated through a series of follow up exams, limited field of view cone beam computed tomography, and periapical radiographs. Additionally, patients will be asked to completed a visual analog scale post surgery for 7 days to track the patients pain response.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary or Mandibular Anterior teeth and premolars #4-13 and #20-29 with a history of failing RCT and a periapical radiolucency will be accepted

Exclusion Criteria:

* Patients with vertical root fractures
* Patients with non-restorable teeth
* Patients with class 3 mobility
* Pregnant
* Smoker
* Systematic disease contraindicating surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in bone deposition using voxel-based imposition | 6 months, 12 months, and 18 months
  From the CBCT images Invivo imaging software (Anatomage, San Jose, CA, USA) will be used to obtain measurements from voxel-based superimposition. The voxel-based imposition is automated by the software to match the voxel grayscale values from the two image volumes. Originally developed by Bazina et al. this analysis method has been demonstrated to show reliable and accurate data. The Linear measurements will be obtained on the cross-section view (sagittal, coronal, and axial) of the periapical lesion on CBCT-1 (6 months) and CBCT-2 (12 months) images.

SECONDARY OUTCOMES:
Healing outcome assessed using clinical and radiographic findings | 6 months, 12 months, and 18 months
  Healing will be assessed by two, board-certified endodontists and a board-certified maxillofacial radiologist. If a consensus cannot be reached, an additional board-certified endodontist will assist in the determination. Healing assessment assisted with 2D imaging will be classified according to Friedmann. These will include healed, healing, or persistent disease. Each will be given a grade of 1-3, one being healed and 3 being persistent disease.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schachman, DMD, Principal Investigator
Locations (1):
- University of Kentucky College of Dentistry Endodontics Division, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time we are undecided if IPD will be shared.

REFERENCES:
- [Background] Miron RJ, Moraschini V, Fujioka-Kobayashi M, Zhang Y, Kawase T, Cosgarea R, Jepsen S, Bishara M, Canullo L, Shirakata Y, Gruber R, Ferenc D, Calasans-Maia MD, Wang HL, Sculean A. Use of platelet-rich fibrin for the treatment of periodontal intrabony defects: a systematic review and meta-analysis. Clin Oral Investig. 2021 May;25(5):2461-2478. doi: 10.1007/s00784-021-03825-8. Epub 2021 Feb 20. PMID 33609186
- [Background] Fan Y, Perez K, Dym H. Clinical Uses of Platelet-Rich Fibrin in Oral and Maxillofacial Surgery. Dent Clin North Am. 2020 Apr;64(2):291-303. doi: 10.1016/j.cden.2019.12.012. Epub 2020 Feb 3. PMID 32111269
- [Background] Mehta N, Gupta A, Aggarwal V, Abraham D, Singh A. Effect of autologous platelet aggregates on the healing outcome of periapical surgery for the management of apicomarginal defects: A systematic review. Saudi Endodontic Journal. 2020 Sep 1;10(3):187- DOI:10.4103/sej.sej_146_19
- [Background] Yan L, Lin J, Yang L, He S, Tan X, Huang D. Clinical Effect Evaluation of Concentrated Growth Factor in Endodontic Microsurgery: A Cross-Sectional Study. J Endod. 2023 Jul;49(7):836-845. doi: 10.1016/j.joen.2023.05.005. Epub 2023 May 12. PMID 37182792
- [Background] Tsesis I, Rosen E, Tamse A, Taschieri S, Del Fabbro M. Effect of guided tissue regeneration on the outcome of surgical endodontic treatment: a systematic review and meta-analysis. J Endod. 2011 Aug;37(8):1039-45. doi: 10.1016/j.joen.2011.05.016. PMID 21763891
- [Background] Pinto D, Marques A, Pereira JF, Palma PJ, Santos JM. Long-Term Prognosis of Endodontic Microsurgery-A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2020 Sep 3;56(9):447. doi: 10.3390/medicina56090447. PMID 32899437
- [Background] Torabinejad M, Corr R, Handysides R, Shabahang S. Outcomes of nonsurgical retreatment and endodontic surgery: a systematic review. J Endod. 2009 Jul;35(7):930-7. doi: 10.1016/j.joen.2009.04.023. PMID 19567310
- [Background] Rud J, Andreasen JO, Jensen JE. Radiographic criteria for the assessment of healing after endodontic surgery. Int J Oral Surg. 1972;1(4):195-214. doi: 10.1016/s0300-9785(72)80013-9. No abstract available. PMID 4199168
- [Background] Gorni FG, Gagliani MM. The outcome of endodontic retreatment: a 2-yr follow-up. J Endod. 2004 Jan;30(1):1-4. doi: 10.1097/00004770-200401000-00001. PMID 14760899
- [Background] Maddalone M, Gagliani M. Periapical endodontic surgery: a 3-year follow-up study. Int Endod J. 2003 Mar;36(3):193-8. doi: 10.1046/j.1365-2591.2003.00642.x. PMID 12657145
- [Background] Setzer FC, Kratchman SI. Present status and future directions: Surgical endodontics. Int Endod J. 2022 Oct;55 Suppl 4:1020-1058. doi: 10.1111/iej.13783. Epub 2022 Jul 4. PMID 35670053